CLINICAL TRIAL: NCT06884020
Title: Estudi De La Desregulació Emocional En Escolars De Dues Etapes Evolutives: Avaluació, Detecció I Intervenció
Brief Title: Emotional Regulation in School and Family: Assessment and Intervention
Acronym: REGUL-EM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, SÍLVIA SEVERINO FANERO, Educational psychologist - Teacher, University Rovira i Virgili
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CEIPSA-2023-TD-0081; DI00036 (Other Grant/Funding Number: Agència de Gestió d'Ajuts Universitaris i Recerca AGAUR)
Record Dates: First submitted 2025-02-27; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Emotional Regulation
Keywords: emotional regulation; emotional education program; pre-school age; School environment; childhood; school-age
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: There are two groups in this project. One group will receive the emotional education intervention first, and when this group and the control group (who did not receive the intervention) complete the post-intervention assessment, the control group will also receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Group 1:
  Pre-assessment: Assessment of emotional regulation, psychological problems and executive functioning through behavioural tests completed by parents and teachers.
  Intervention: Participants receive a weekly emotional education program (8 sessions of 45 minutes each, plus an additional 1-hour session with the family in the middle of the program).
  Intervention facilitator: A doctoral student (psychologist and teacher) conducts the sessions.
  Participants: The program is offered to the entire group of 5-year-old preschool children (I5), regardless of their pre-assessment results, with the informed consent of parents or guardians.
  Location: The intervention will be delivered in the early childhood education classroom.
  Post-intervention evaluation: Conducted both in the short term (immediately after the end of the program) and in the medium to long term (4-5 months after the end of the program).
  Interventions: Behavioral: EMOTIONAL REGULATION PROGRAMME
- Control group (No Intervention): Group 2:
  Pre-assessment: Similar to group 1, assessment of emotional regulation, psychological problems and executive functioning through behavioural tests completed by parents and teachers.
  Intervention: This group will not receive the emotional education program during the initial phase of the study.
  Participants: The entire group of 5-year-old preschool children (I5), with the informed consent of parents or guardians.
  Post-assessment:
  Short-term evaluation: Conducted at the same time as Group 1, immediately after the end of the intervention program for the experimental group.
  Medium to long-term evaluation: Conducted at the same time as Group 1, 4-5 months after the end of the intervention programme for the experimental group. The control group will not receive the intervention until after this evaluation.
  Intervention facilitator: A doctoral student (psychologist and trained teacher).
  Location: The intervention will be delivered in the early childhood education classroom

INTERVENTIONS:
Behavioral: EMOTIONAL REGULATION PROGRAMME — This programme works on early identification and implementation of strategies to improve self-awareness and facilitate children's emotions.
  This intervention is designed to be delivered in the educational setting by the tutor in the form of a learning situation with 8 sessions plus 1 family session.
  The topics covered are:
  * Embarking on an emotional journey
  * Recognising our emotions
  * Emotions have a voice
  * Identifying different emotions
  * How do I make decisions?
  * Emotion, action, and consequence
  * Learning to self-regulate
  * Celebrating our learning
  Arms: Intervention group

SUMMARY:
This project aims to investigate children's difficulties with emotional regulation in the school environment, to develop an early intervention programme for preschool children (5 years old) and their families, and to explore the relationship between emotional regulation and various risk and protective factors, including variables such as gender, age, socio-economic context, parenting styles, social skills and academic performance. Data analysis will facilitate the adaptation of the intervention to the needs of the school population.

Methodologically, the project will adopt a quasi-experimental design with control and experimental groups, using a convenience sample drawn from two schools in Tarragona. This design will make it possible to compare the effectiveness of the programme in improving children's emotional skills.

DETAILED DESCRIPTION:
Emotional regulation skills refer to the way individuals manage their emotional experiences, representing a complex and essential process acquired throughout development. This process is influenced by both neurobiological and social-contextual factors. Acquiring the ability to regulate emotions is fundamental to human functioning and adjustment. Scientific evidence indicates that strong emotional regulation skills are significantly associated with higher levels of social competence, better social relationships, improved academic performance, and greater adaptation to school environment demands, as well as higher resilience levels, among other benefits. Conversely, difficulties in emotional regulation, the inability or limited ability to modulate emotional responses, have been linked to the presence of psychopathological and health problems.

Regarding emotional regulation across the lifespan, Bowlby's attachment theory, in conjunction with Hoffman's Circle of Security, posits that the early years of life are crucial for the initial learning of emotions through primary caregivers. The ability to regulate emotions effectively is shaped by the interactions and modulations a child experiences in their early years with their primary caregivers, as well as through observation and interaction with family members and close acquaintances. Consequently, aspects such as emotional bonds, including those with teachers, and parenting styles are highly relevant. In fact, parental self-regulation, referring to parents' ability to regulate their own emotions, directly interacts with the co-regulation of their children. Co-regulation is understood as the mechanism enabling mutual emotional regulation between individuals. As children and adolescents develop, they acquire more coping strategies and become increasingly capable of attending to and reflecting on their own emotional states and those of others. Cognitive development and brain maturation further enhance their regulatory capacity, making it more effective and adaptive. However, some studies suggest that during mid-adolescence, individuals tend to exhibit fewer adaptive regulation strategies, possibly due to increased parent-child conflicts or heightened emotional difficulties characteristic of this developmental stage. Thus, emotional regulation difficulties are considered a transdiagnostic factor associated with nearly all forms of psychopathology in adolescents.

The prevalence of emotional symptoms and disorders such as anxiety and depression is high in children and adolescents, underscoring the need for prevention and intervention efforts focused on enhancing emotional skills from early developmental stages. These interventions should not be confined solely to the family or social environment of children and adolescents. Various researchers, from both theoretical and practical perspectives, emphasize the importance of integrating emotional education within educational institutions.

Intervention programs designed to strengthen emotional regulation skills generally follow two main approaches. One focuses on working with families and children from the age of three, coinciding with the start of schooling and the expansion of social relations beyond the family. The other consists of programs implemented in classrooms, targeting primary and secondary education. Notably, emotional intelligence programs in secondary education emphasize conflict resolution and classroom coexistence. Programs such as Conflict Mediation and CONVES: Program to Improve School Coexistence indicate that secondary education initiatives outnumber those in primary education by a ratio of two to one and exceed early childhood programs fourfold, highlighting the need for research and development efforts at the earliest educational stages.

Given the growing interest in fostering emotional well-being in classrooms and recognizing teachers as facilitators of emotional learning, this approach enhances students' self-awareness and decision-making skills, goal attainment, and conflict resolution abilities. This paradigm shift has led to an increased emphasis on incorporating learning experiences that support children's emotional well-being within the education system. This is evident in the recent implementation of DECRET 175/2022, de 27 de September, which governs basic education curricula and emphasizes the importance of holistic student development through six vectors, particularly the sixth, named Emotional Well-being.

Further research is needed on emotional regulation, incorporating assessments from multiple informants and across different developmental stages. Additionally, a deeper exploration of genetic and environmental factors influencing children's emotional regulation abilities in the current social context is necessary. Moreover, there is a pressing need for tailored programs for earlier developmental stages, designed for both children and their families. Advancing research in this domain is essential, as emotional competence is a crucial aspect of human development throughout the lifespan.

Methodology The primary objective of this project is to assess emotional regulation difficulties in children at different educational levels within the school environment and to design an early intervention program (targeted at preschool-aged children and their families) for implementation and follow-up in the short, medium, and long term. Furthermore, the study aims to examine the relationship between emotional regulation and various risk and protective factors, considering multiple sociodemographic and educational variables. Emotional regulation difficulties will be analysed concerning factors such as gender, age/educational level, ethnicity, and family socioeconomic status, as well as parenting styles, attachment bonds, cognitive abilities, social skills, emotional and/or behavioural strengths and weaknesses, and academic aspects such as performance or learning difficulties. The collected data will facilitate the adaptation of preventive interventions to the target school population.

The project will involve conducting a comprehensive and specific assessment based on participants' developmental stages. Information will be collected from different informants: teachers, families, and self-reports from pupils (from age eight onwards). In the second phase, a universal early preventive intervention program will be designed and implemented, targeting children and families in Year 1, followed by a subsequent re-evaluation. Teachers, children, and families from The British School of Costa Daurada, a private school managed by Servei d'Atenció als Infants Tarragona SL, will participate. The sample may be expanded to include participants from other schools in the province of Tarragona to enable a comparative study.

The phases of the project are as follows: Phase 0: Project preparation, documentation, and obtaining necessary administrative permits, with approval from the Ethics Committee of Rovira i Virgili University. Phase 1: Explanation of the project to families and obtaining informed consent. Implementation of the study's assessment protocol (pre-intervention assessment), test correction, and data management and analysis. Phase 2: Design and creation of the intervention program and preparation of necessary materials. Implementation of the intervention program at the early childhood education stage (with an experimental and a control group, as detailed in the Study Design section). Phase 3: Post-intervention assessment. Phase 4: Follow-up session on the intervention 4-6 months afterward. Phase 5: Post-intervention assessment 7-9 months later. Phase 6: Data analysis and dissemination of results.

The study employs validated instruments to assess emotional regulation, behavioural functioning, and parental stress. These include the Cognitive Emotion Regulation Questionnaire and its pre-adolescent version, the Behavioural Assessment System for Children-3, and the Behaviour Rating Inventory of Executive Function. Parenting-related factors are measured using the Parenting Stress Index and The Parenting Scale. Additionally, a custom questionnaire has been developed to collect sociodemographic and educational data.

ELIGIBILITY:
Student of Early Childhood Education

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Emotional Self-Control (BASC-3 Scores) | Baseline (Week 5), post-intervention (Week 15 and Week 45).
  Assessment of emotional self-control using the BASC-3, completed by parents/guardians and school staff. Higher scores indicate lower emotional self-control and greater difficulty in managing emotions effectively.
  BASC-3 scores range from 0 to 120, where higher scores reflect greater difficulties in emotional self-control.
Emotional Regulation (BRIEF-P Scores) | Baseline (Week 5), post-intervention (Week 15 and Week 45).
  Assessment of emotional regulation using the BRIEF-P, completed by parents/guardians and school staff. Higher scores indicate greater emotional dysregulation, reflecting difficulties in managing and modulating emotional responses effectively.
  BRIEF-P scores range from 30 to 90, where higher scores reflect greater emotional dysregulation.

SECONDARY OUTCOMES:
Behavioral and Emotional Problems (BASC-3 Scores) | Baseline (Week 5 of the school year) Post-intervention (Week 15 and Week 45 of the school year) Follow-up (Up to 1 year after study completion)
  Assessment of behavioural and emotional difficulties using the BASC-3, completed by parents/legal guardians and school staff. This measure evaluates emotional symptoms, conduct issues, hyperactivity/inattention, peer relationship difficulties, and overall behavioural functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Josefa Dra. Canals, Full Professor, Study Director — University Rovira i Virgili
Locations (1):
- Universitat Rovira i Virgili, Tarragona, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The decision will be made on the basis of the URV's institutional policy and ethical requirements.